CLINICAL TRIAL: NCT02503657
Title: A Randomized, Placebo-Controlled, Double-Blind Six Month Study Followed by an Open-Label Extension Phase to Evaluate the Efficacy, Safety and Tolerability of MN-001 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Safety, Tolerability, and Efficacy of MN-001 (Tipelukast) in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN-001-IPF-201
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; IPF
Keywords: tipelukast; IPF; fibrosis; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — 4-(6-acetyl-3-(3-(4-acetyl-3-hydroxy-2-propylphenylthio)propoxy)-2-propylphenoxy)butyric acid

STUDY DESIGN:
Intervention Model Description: This study evaluated the efficacy, safety, and tolerability of MN-001 in male and female patients aged 21 to 80 years, inclusive, with moderate-to-severe idiopathic pulmonary fibrosis (IPF). Fifteen (15) participants received MN-001 750 mg or a matching placebo twice daily for 26 weeks in a 2:1 (MN-001:Placebo) ratio. The study consisted of a Screening period (up to 3 months before baseline), a 26-week double-blind treatment (DBT) period, a 26-week open-label (OL) treatment period, and a follow-up visit (within 4 weeks after the last dose). Efficacy results are reported only for the DBT period. Safety findings are reported from Baseline (Day 1 of MN-001 or placebo treatment) to the end of the Open-Label period (52 weeks total).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The double-blind period is masked by the participants, care provider, investigator, and outcomes assessor.
Oversight: Data Monitoring Committee: No

ARMS (2):
- MN-001 in Double-blind period for 26 weeks, then MN-001 in Open-Label period for 26 weeks (Experimental): MN-001 750 mg twice a day during the double-blind period (26 weeks) and MN-001 750 mg twice a day during the open-label period for 26 weeks. The arm title is shortened to MN-001/MN-001 for all results sections.
  Interventions: Drug: MN-001
- Placebo during Double-blind period for 26 weeks, then MN-001 in Open-Label period for 26 weeks (Placebo Comparator): Placebo twice a day during the double-blind period for 26 weeks and MN-001 750 mg twice daily during the open-label period for 26 weeks. The arm title is shortened to Placebo/MN-001 for all results sections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MN-001 — A novel, orally bioavailable small molecule compound that demonstrates anti-inflammatory and anti-fibrotic activity
  Other Names: Tipelukast
  Arms: MN-001 in Double-blind period for 26 weeks, then MN-001 in Open-Label period for 26 weeks
Drug: Placebo — Excipients of MN-001/tipelukast
  Arms: Placebo during Double-blind period for 26 weeks, then MN-001 in Open-Label period for 26 weeks

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 6-month study followed by a 6-month open-label extension phase to evaluate the efficacy, safety, and tolerability of MN-001 in patients diagnosed with moderate to severe idiopathic pulmonary fibrosis (IPF). Participants were randomly assigned to receive MN-001 or matching placebo twice daily over a 26-week period. A total of 15 participants were enrolled.

DETAILED DESCRIPTION:
This study was a single-center, randomized (2:1), placebo-controlled, double-blind, 6-month study followed by a 6-month open-label extension (OLE) phase in patients with moderate to severe IPF. Major inclusion criteria: physician diagnosed IPF (ATS Guidelines, 2011), males and females aged 21 to 80 years, GAP Stage II-III; on no anti-fibrotic treatment. Patients on stable dose of nintedanib for at least 3 months prior to the study were allowed.

The study consisted of a Screening Phase (up to 3 months prior to Day1), a 26- week Double-Blind Treatment (DBT) period, a 26-week Open-Label Extension (OLE) period, and a Follow-up / End of Study Visit (within 4 weeks of the last dose taken).

A total of 15 patients were enrolled in the study. During the DBT period, participants were randomly assigned to receive MN-001 750 mg twice daily or a matching placebo in a 2:1 ratio (MN-001: placebo) for 26 weeks. During the OLE period, all participants received MN-001 750 mg twice daily for 26 weeks. Taken together, participants (n=15) received either MN-001 50 mg twice daily for 12 months (MN-001/MN-001) or matching placebo for 6 months and MN-001 750 mg twice daily for 6 months (Placebo/MN-001).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ages 21 to 80, inclusive
* Presence of IPF confirmed per ATS criteria (2011)
* Presence of moderate to severe disease, stage II-III defined by GAP index (Gender, Age and Physiology)
* Subjects who are currently treated with OFEV™/Nintedanib should be on a stable dose for at least 3 months prior to initiation of the study drug.
* Females of child-bearing potential must have a negative serum ß-hCG (human chorionic gonadotropin) at screening and must be willing to use appropriate contraception (as defined by the investigator) for the duration of study treatment and 30 days after the last dose of study treatment.
* Males should practice contraception for the duration of study treatment and 30 days after the last dose of study treatment as follows: condom use and contraception by female partner.
* Subject is in stable condition on the basis of medical history, physical examination, and laboratory screening, as determined by the investigator.
* Subject is willing and able to comply with the protocol assessments and visits, in the opinion of the study nurse/coordinator and the Investigator.
* Written informed consent is obtained prior to participating the study.

Exclusion Criteria:

* Expected to receive a lung transplant within 1 year from the start of the Treatment Phase or on a lung transplant waiting list at the start of the Treatment Phase.
* Known explanation for interstitial lung disease
* Subjects on OFEV™/Nintedanib with a dose interruption due to significant adverse events within 6 weeks of screening visits.
* Ongoing IPF treatments with investigational therapy
* Ongoing IPF treatments with Esbriet® (Pirfenidone)
* Immunosuppressants (i.e., Mycophenolate, Imuran, Cyclophosphamide), and cytokine modulating agents within 1 month of Screening Visit and throughout the study
* Use of antibiotics and systemic steroids due to IPF exacerbation within 1 month of Screening Visit
* Clinically significant cardiovascular disease, including myocardial infarct within last 6 months, unstable ischemic heart disease, congestive heart failure or angina
* Resting pulse < 50 bpm, SA (sinoatrial) or AV (atrioventricular) block, uncontrolled hypertension, or QTcF (QT interval corrected using the Fridericia formula) > 450 ms
* Immune system disease
* Any significant laboratory abnormality which, in the opinion of the Investigator, may put the subject at risk
* History of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* History or evidence of drug or alcohol abuse
* History of HIV (human immunodeficiency virus) or other active infection.
* Currently has a clinically significant medical condition including the following: neurological, psychiatric, immunological, metabolic, hepatic, hematological, pulmonary (other than IPF) , cardiovascular (including uncontrolled hypertension), gastrointestinal, urological disorder, or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if, in the judgment of the Investigator, they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted.

* CYP2C8 (cytochrome P450 isoenzyme C28) and CYP2C9 (cytochrome P450 isoenzyme C29) substrates with narrow therapeutic indices (i.e. paclitaxel, phenytoin and S-warfarin) within 14 days of Screening Visit and throughout the study.
* Beta blockers within 14 days of Screening Visit and throughout the study
* Macrolide or quinolone class antibiotics within 14 days of Screening Visit and throughout the study.
* Poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator.
* Currently participating, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent.
* Unwilling or unable to conduct Spirometry (Vital Capacity) test.
* Unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator, or is planning to relocate during the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Bascom, MD, Principal Investigator — PSU Research, Department of Medicine
Locations (1):
- Penn State University College of Medicine, Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site.
Pre-assignment Details: In the double-blind period, participants were randomly assigned to receive MN-001 or placebo in a 2:1 ratio, meaning that 10 participants received MN-001 and 5 participants received placebo. In the Open-label period, all 15 participants who completed the double-blind period received MN-001.
Groups:
- MN-001/MN-001: MN-001 (tipelukast) 750 mg tablet by mouth twice daily for 26 weeks.
  MN-001: A novel, orally bioavailable small molecule compound that demonstrates anti-inflammatory and anti-fibrotic activity
- Placebo/MN-001: Matching placebo twice a day for 26 weeks.
  Matching Placebo: Excipients of MN-001/tipelukast
Period: Double-blind Period
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0
Period: Open-label Period
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Started | 10 | 5
Completed | 10 | 4
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MN-001/MN-001 | Placebo/MN-001 | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (5.8) | 66.2 (9.6) | 69.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Forced Vital Capacity for 26 Weeks
Description: Predicted forced vital capacity (FVC) is a reference value for lung function based on your age, height, sex, and ethnicity measured by a spirometer and is an established method of pulmonary function. FVC is the volume of air that can be forcibly blown out after full inspiration, measured in liters (L).
Time Frame: Baseline and Week 26 at the end of Double-blind treatment period.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Placebo/MN-001: Matching placebo twice daily for 26 weeks.
  Matching Placebo: Excipients of MN-001/tipelukast
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 10 | 5
Liters | -0.177 (0.270) | -0.025 (0.233)

2. Primary Outcome: Percent Change in Forced Vital Capacity From Baseline to Week 26
Description: FVC is the volume of air that can be forcibly blown out after full inspiration, measured in liters (L). The mean relative change was calculated as 100*[FVC (L) at Week 26 - FVC (L) at baseline].
Time Frame: Baseline, and Week 26 at the endpoint of the Double-blind treatment period.
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 9 | 4
percent of change | -7.22 (10.02) | -0.33 (10.45)

3. Primary Outcome: Absolute Change From Baseline in Forced Vital Capacity (% Predicted)
Description: FVC(%pred.) refers to the expected FVC for a healthy individual with the same age, sex, height, and weight. The actual FVC result is then expressed as a percentage of this predicted value; values of 80% or higher are generally considered normal and indicate no significant impairment.
Time Frame: Baseline and Week 26 at the end of Double-blind treatment period.
Measure: Mean (Standard Deviation); unit: percent predicted normal volume
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 9 | 4
percent predicted normal volume | -5.60 (7.00) | -0.56 (5.49)

4. Primary Outcome: Relative Change From Baseline in Percent Predicted Forced Vital Capacity From Baseline to Week 26
Description: FVC (%pred/) refers to the expected FVC for a healthy individual with the same age, sex, height, and weight. The actual FVC result is then expressed as a percentage of this predicted value; values of 80% or higher are generally considered normal and indicate no significant impairment. Relative change is measured as percent (%) change from FVC (%pred.).
Time Frame: Baseline and Week 26 at the end of Double-blind treatment period.
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 9 | 4
percent of change | -7.22 (10.02) | -0.33 (10.45)

5. Primary Outcome: Semiannual Rate of Decline of Disease Activity Based on Forced Vital Capacity
Description: The semiannual rates of change in FVC, measured in liters, were estimated using simple linear regression, with time measured in half-years.
Time Frame: Baseline and Week 26 at the end of Double-blind treatment period.
Measure: Mean (Standard Deviation); unit: Liters per year
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 10 | 5
Liters per year | -0.1776 (0.2501) | 0.0131 (0.2118)

6. Secondary Outcome: Number of Participants With Treatment-related Serious Adverse Events.
Description: Treatment-related serious adverse events (TRSAEs) are defined as possibly related, probably related, or related to MN-001 treatment.
Time Frame: Baseline, and Week 26 at the endpoint of the Double-blind treatment period
Population: (TRSAEs) are reported by treatment period: 1) Double-blind MN-001 treatment, 2) Double-blind Placebo treatment, and 3) Open-Label MN-001 treatment for all participants, regardless of assignment in the Double-blind period.
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind MN-001: MN-001 (tipelukast) 750 mg tablet by mouth twice daily for 26 weeks (n=10)
  MN-001: A novel, orally bioavailable small molecule compound that demonstrates anti-inflammatory and anti-fibrotic activity
- Double-blind Placebo: Matching placebo twice daily for 26 weeks (n=5)
  Matching Placebo: Excipients of MN-001/tipelukast
- OLE MN-001: MN-001 (tipelukast) 750 mg tablet by mouth twice daily for 26 weeks (n=15).
  MN-001: A novel, orally bioavailable small molecule compound that demonstrates anti-inflammatory and anti-fibrotic activity
Arm/Group | Double-blind MN-001 | Double-blind Placebo | OLE MN-001
Number analyzed (Participants) | 10 | 5 | 15
Participants | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline on Disease Activity Based on Modified Medical Research Council Dyspnea Score
Description: The Modified Medical Research Council Dyspnea Score is a simple grading system widely used in the assessment of dyspnea (difficulty breathing) in chronic respiratory diseases, such as IPF. The breathlessness scale comprises five statements that cover respiratory disability from 0 (zero) to 4, in which 0 = not troubled by breathlessness, except on strenuous exercise, 1= shortness of breath when hurrying on the level or walking up a slight hill, 2 = walks slower than people of the same age or has to stop for breath when walking at own pace on level ground, 3 = stops for breath after walking just 100 meters (100 yards) or after a few minutes, and 4 = too breathless to leave the house or breathless when dressing or undressing. A higher score corresponds to greater difficult in breathing.
Time Frame: Baseline, and Week 26 at the endpoint of the Double-blind treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 9 | 4
score on a scale | 0.8 (0.7) | 0.5 (1.0)

8. Secondary Outcome: Change From Baseline on Quality of Life (QOL) Measured by A Tool to Assess Quality of Life in Idiopathic Pulmonary Fibrosis
Description: The A Tool to Assess Quality of Life in Idiopathic Pulmonary Fibrosis score is a quality-of-life questionnaire that has 13 domains (cough, dyspnea, forethought, sleep, mortality, exhaustion, emotional well-being, social participation, finances, independence, sexual health, relationships, therapy). The domain scores and the Total score from these domain scores are calculated by summation. Higher scores correspond to greater impairment. The Total score ranges from 74 to 370.
Time Frame: Baseline, and Week 26 at the endpoint of the Double-blind treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 9 | 4
score on a scale | 16.8 (55.7) | -5.3 (28.0)

9. Secondary Outcome: Frequency of Worsening IPF
Description: The number of participants who experienced worsening in IPF. Worsening of IPF is defined as acute IPF exacerbation, hospitalization due to respiratory symptoms, IPF-related fatal events, and/or lung transplantation.
Time Frame: Baseline, and Week 26 at the endpoint of the Double-blind treatment period
Measure: Number; unit: number of participants
Arm/Group | MN-001/MN-001 | Placebo/MN-001
Number analyzed (Participants) | 10 | 5
number of participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 26 weeks in the double-blind treatment period, 26 weeks in the open-label period
Groups:
- Open Label MN-001/Former Placebo: MN-001 (tipelukast) 750 mg tablet by mouth twice daily for 26 weeks (n=15).
  MN-001: A novel, orally bioavailable small molecule compound that demonstrates anti-inflammatory and anti-fibrotic activity
Arm/Group | Double-blind MN-001 | Double-blind Placebo | Open Label MN-001/Former Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/5 | 3/15
Other Adverse Events (participants affected / at risk) | 10/10 | 5/5 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MN-001 (N=10) | Double-blind Placebo (N=5) | Open Label MN-001/Former Placebo (N=15)
Femur fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MN-001 (N=10) | Double-blind Placebo (N=5) | Open Label MN-001/Former Placebo (N=15)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eosinophelia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Polllakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02503657/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02503657/SAP_001.pdf